CLINICAL TRIAL: NCT01050517
Title: Gaps in Helminth Control: Safety and Efficacy of Drug Combinations Against Triple Infections
Brief Title: Safety and Efficacy of Drug Combinations Against Triple Infections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DBL -Institute for Health Research and Development (Other)
Responsible Party: Harriet Namwanje, Vector Control Division, MOH
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AO.UGA.TRIPLE; DBL-CHRD
Record Dates: First submitted 2008-01-23; First posted 2010-01-15 (Estimated); Last update posted 2010-01-15 (Estimated); Status verified 2010-01

CONDITIONS: Parasitic Diseases
MeSH Terms: conditions — Parasitic Diseases | interventions — Albendazole; Ivermectin; Praziquantel

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): albendazole + ivermectin + praziquantel
  Interventions: Drug: albendazole + ivermectin + praziquantel
- 2 (Placebo Comparator): albendazole + ivermectin + (1 week later) praziquantel
  Interventions: Drug: albendazole + ivermectin + (1 week later) praziquantel

INTERVENTIONS:
Drug: albendazole + ivermectin + praziquantel — albendazole (400 mg one dose) + ivermectin 200 microgram/kg body weight) + praziquantel (40 mg/kg)
  Arms: 1
Drug: albendazole + ivermectin + (1 week later) praziquantel — albendazole (400 mg one dose) + ivermectin (200 microgram/kg body weight) + (1 week later) praziquantel (40 mg/kg)
  Arms: 2

SUMMARY:
This randomised, controlled, double blinded clinical study investigates the safety and efficacy of the combination of albendazole, ivermectin and praziquantel in the treatment of children aged 5-18 years co-infected with lymphatic filariasis, schistosomiasis and soil-transmitted helminthiasis.

ELIGIBILITY:
Inclusion Criteria:

* Those who will be in class one to six by the time of study
* Aged 5-18 years and found infected with either SCH, any STH or LF for treatment groups 1,2 or 3 or infected with both SCH and LF for treatment group 4 and infected with all the three for treatment group 5
* Who are willing and consent and whose parents will consent, will be included in the study.

Exclusion Criteria:

* Those with acute and chronic diseases other than the targeted infections and those with a history of any serious adverse drug reactions will not be included in the study.
* Children with total bilirubin > 50µmol/L and ALAT (Alanine transferase) > 70IU/L will not qualify for recruitment.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 250 (Estimated)
Dates: Start 2007-10; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
adverse reactions | 6 weeks

SECONDARY OUTCOMES:
Efficacy of treatment | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Vector Control Division, Kampala, Uganda

REFERENCES:
- [Derived] Namwanje H, Kabatereine N, Olsen A. A randomised controlled clinical trial on the safety of co-administration of albendazole, ivermectin and praziquantel in infected schoolchildren in Uganda. Trans R Soc Trop Med Hyg. 2011 Apr;105(4):181-8. doi: 10.1016/j.trstmh.2010.11.012. Epub 2011 Feb 25. PMID 21353271